CLINICAL TRIAL: NCT03801928
Title: OBSERVATIONAL, REAL WORLD STUDY OF INFLECTRA IN PATIENTS WITH INFLAMMATORY BOWEL DISEASE (IBD) IN THE UNITED STATES AND CANADA
Brief Title: Observational, Real World Study Of Inflectra In Patients With Inflammatory Bowel Disease
Acronym: ONWARD
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1231006; ONWARD (Other: Alias Study Number)
Record Dates: First submitted 2018-12-11; First posted 2019-01-14 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn's Disease (CD); Ulcerative Colitis (UC)
Keywords: Inflectra; Remicade
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ulcerative Colitis: Group treated with Inflectra for Ulcerative Colitis
  Interventions: Drug: Inflectra
- Crohn's Disease: Group treated with Inflectra for Crohn's Disease
  Interventions: Drug: Inflectra

INTERVENTIONS:
Drug: Inflectra — The study plans to recruit 300 subjects in the United States and Canada initiating or switching to treatment with INFLECTRA over an 8 month period. The decision to start INFLECTRA will be entirely a clinical decision made by the participating physician irrespective of this study.
  Other Names: Infliximab

SUMMARY:
This is a prospective, observational, multicenter study conducted in adult patients with ulcerative colitis (UC) or Crohn's disease (CD). The study plans to recruit 300 subjects in the United States and Canada in which the participating physician has decided to treat with INFLECTRA. The study will evaluate treatment patterns, adherence, disease activity, remission status, relapse status, treatment satisfaction, and healthcare resource utilization. Patient outcomes will be assessed at four time points (quarterly) for approximately 52 weeks after the decision to initiate treatment with INFLECTRA.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for inclusion in the study:

1. Patients with confirmed diagnosis of Ulcerative Colitis or Crohn's Disease.
2. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
3. Patient eligible to receive INFLECTRA for the treatment of their disease per approved drug label (patients with fistula, or stoma are eligible).

Exclusion Criteria:

-Patients meeting any of the following criteria will not be included in the study:

1. Patient previously failed treatment with REMICADE or INFLECTRA/CT P13.
2. Any reported contraindications for INFLECTRA/CT P13 or REMICADE.
3. Known hypersensitivity (including severe, acute infusion reactions) to infliximab, its excipients or other murine proteins, at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients are planned to be enrolled from approximately 30 40 physician clinics. Enrollment is planned to be competitive, but an upper limit of 20 patients per site per cohort will be applied to maintain the generalizability of the study. This is an observational study; therefore the decision to treat a patient with INFLECTRA must be made prior to a decision to enroll them in this study. Patients are eligible to participate if they have:
  * Initiated therapy with INFLECTRA as their first biologic;
  * Switched to INFLECTRA while in remission on a stable dose of REMICADE; or,
  * Switched to INFLECTRA from another biologic, due to non responsiveness, intolerance, or other reasons.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (11):
  - San Diego Clinical Trials, San Diego, California
  - Medical Research Center Of Connecticut, LLC, Hamden, Connecticut
  - Suncoast Research Group, LLC, Miami, Florida
  - Illinois Gastroenterology Group, Gurnee, Illinois
  - Indiana University Health Division of Gastroenterology/Hepatology, Indianapolis, Indiana
  - Gastro Center of Maryland, Columbia, Maryland
  - Infusion Associates N.E., Grand Rapids, Michigan
  - Trinity Health Center Medical Arts, Minot, North Dakota
  - Dayton Gastroenterology, Inc., Beavercreek, Ohio
  - Paramount Medical Research & consulting, LLC, Middleburg Heights, Ohio
  - The Vancouver Clinic Research, Vancouver, Washington
- Canada (4):
  - Aspen Woods Clinic, Calgary, Alberta
  - Brennan Walters Professional Corporation, Edmonton, Alberta
  - Fraser Clinical Trials, New Westminster, British Columbia
  - Montreal IBD Center (CMIIM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Abraham B, Eksteen B, Nedd K, Kale H, Patel D, Stephens J, Shelbaya A, Chambers R, Soonasra A. Impact of Infliximab-dyyb (Infliximab Biosimilar) on Clinical and Patient-Reported Outcomes: 1-Year Follow-up Results from an Observational Real-World Study Among Patients with Inflammatory Bowel Disease in the US and Canada (the ONWARD Study). Adv Ther. 2022 May;39(5):2109-2127. doi: 10.1007/s12325-022-02104-6. Epub 2022 Mar 16. PMID 35296993
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1231006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included had inflammatory bowel disease (IBD), with a confirmed diagnosis of ulcerative colitis (UC) or Crohn's disease (CD): 1) those who newly initiated therapy with Inflectra as their first biologic, 2) transitioned to Inflectra from Remicade, 3) switched to Inflectra from other biologics. Total 118 participants were enrolled and assessed for eligibility. Out of 118, only 115 participants received Inflectra and were eligible to be included in the study.
Pre-assignment Details: Participants initiated or switched to Inflectra in a real-world setting and it was a decision made by physician irrespective of this study. Inflectra dose was per summary of product characteristics as determined by physician, for every 8 weeks. Participants were observed and evaluated prospectively at 4 study visits (visit 1= Day 1, visit 2= Day 90, visit 3= Day 180, visit 4= Day 365; all visits were from first dose of Inflectra) for approximately (approx.) 1 year after treatment with Inflectra.
Groups:
- UC: New Inflectra: Participants included in this arm had a confirmed diagnosis of UC, with no previous biologics use and who in a real world setting received intravenous infusions of Inflectra as their first biologic.
- UC: Inflectra After Remicade: Participants included in this arm had a confirmed diagnosis of UC, who had previous treatment with stable dose of Remicade and who in a real world setting received intravenous infusions of Inflectra after transition from Remicade.
- UC: Inflectra After Other Biologics: Participants included in this arm had a confirmed diagnosis of UC, who had previous treatment with stable dose of other biologics and who in a real world setting received intravenous infusions of Inflectra after switching from other biologics.
- CD: New Inflectra: Participants included in this arm had a confirmed diagnosis of CD, with no previous biologics use and who in a real world setting received intravenous infusions of Inflectra as their first biologic.
- CD: Inflectra After Remicade: Participants included in this arm had a confirmed diagnosis of CD, who had previous treatment with stable dose of Remicade and who in a real world setting received intravenous infusions of Inflectra after transition from Remicade.
- CD: Inflectra After Other Biologics: Participants included in this arm had a confirmed diagnosis of CD, who had previous treatment with stable dose of other biologics and who in a real world setting received intravenous infusions of Inflectra after switching from other biologics.
Period: Overall Study
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Started | 18 | 21 | 9 | 21 | 36 | 10
Completed | 12 | 18 | 4 | 13 | 32 | 5
Not Completed | 6 | 3 | 5 | 8 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 1 | 4 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who signed the informed consent and met the study inclusion/exclusion criteria in the study design, or the subgroups as following: those who newly initiated Inflectra, transitioned to Inflectra from Remicade or switched to Inflectra from other biologics.
Groups:
- Total: Total of all reporting groups
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics | Total
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10 | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.94 (17.72) | 41.76 (12.68) | 51.67 (16.39) | 46.86 (17.98) | 43.40 (17.02) | 39.00 (14.51) | 44.25 (16.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 6 | 8 | 19 | 6 | 59
  Male | 10 | 9 | 3 | 13 | 17 | 4 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 1 | 1 | 0 | 3
  Black or African American | 0 | 1 | 1 | 2 | 3 | 1 | 8
  White or Caucasian American | 16 | 20 | 6 | 18 | 31 | 9 | 100
  Other | 2 | 0 | 1 | 0 | 1 | 0 | 4
Insurance Plan Coverage [Count of Participants; unit: Participants] — Number of participants were classified on the basis of insurance plan coverage they had.
  Participants
    Canada Medicare | 4 | 0 | 4 | 4 | 0 | 4 | 16
    Health Maintenance Organization (HMO) | 2 | 18 | 0 | 2 | 22 | 2 | 46
    Medicare/Medicaid | 3 | 3 | 3 | 6 | 9 | 1 | 25
    Point of Service Plan (POS) | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Preferred Provider Organization (PPO) | 9 | 0 | 2 | 9 | 4 | 2 | 26
    Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
Surgical History [Count of Participants; unit: Participants] — Number of participants who had undergone previous IBD related surgeries were reported.
  Participants | 0 | 2 | 0 | 4 | 15 | 3 | 24
Disease Duration [Mean (Standard Deviation); unit: Years] — Duration of IBD in years reported.
  Years | 5.96 (6.40) | 8.88 (8.86) | 10.00 (9.11) | 5.89 (6.30) | 10.59 (10.28) | 7.22 (7.45) | 8.26 (8.47)
Medication History [Count of Participants; unit: Participants] — Number of participants who previously received anti-tumor necrosis factor (TNF) disease related medications were reported.
  Participants | 0 | 21 | 9 | 1 | 36 | 9 | 76
Concomitant Medication Usage [Count of Participants; unit: Participants] — Number of participants who previously received concomitant medications (medications other than for IBD) were reported.
  Participants | 18 | 14 | 7 | 18 | 16 | 9 | 82

OUTCOME MEASURES:

1. Primary Outcome: Average Dose of Inflectra at Visit 1
Time Frame: Visit 1= Day 1
Population: The full analysis set included all participants who signed the informed consent and met the study inclusion/exclusion criteria in the study design, or the subgroups as following: those who newly initiated Inflectra, transitioned to Inflectra from Remicade or switched to Inflectra from other biologics. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 35 | 10
milligram | 457.28 (184.03) | 585.71 (305.43) | 579.44 (193.69) | 449.76 (102.33) | 521.83 (274.76) | 534.90 (171.15)

2. Primary Outcome: Average Dose of Inflectra at Visit 2
Time Frame: Visit 2= Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 17 | 17 | 8 | 20 | 32 | 8
milligram | 491.66 (201.43) | 535.29 (259.67) | 662.36 (194.54) | 491.62 (172.95) | 506.97 (236.03) | 575.00 (210.76)

3. Primary Outcome: Average Dose of Inflectra at Visit 3
Time Frame: Visit 3= Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 16 | 16 | 5 | 15 | 30 | 5
milligram | 556.34 (216.05) | 531.25 (270.11) | 647.67 (328.73) | 517.87 (162.06) | 544.40 (233.21) | 621.00 (230.55)

4. Primary Outcome: Average Dose of Inflectra at Visit 4
Time Frame: Visit 4= Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 9 | 15 | 2 | 9 | 26 | 4
milligram | 409.28 (216.59) | 552.00 (270.43) | 450.00 (70.71) | 536.12 (216.39) | 553.20 (238.22) | 610.15 (229.08)

5. Primary Outcome: Mean Number of Inflectra Infusions at Visit 1
Time Frame: Visit 1= Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 35 | 10
infusions | 1.56 (0.62) | 1.00 (0.00) | 1.44 (0.53) | 1.43 (0.51) | 1.11 (0.32) | 1.70 (0.67)

6. Primary Outcome: Mean Number of Inflectra Infusions at Visit 2
Time Frame: Visit 2= Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 17 | 17 | 8 | 20 | 32 | 8
infusions | 2.06 (0.75) | 1.76 (0.44) | 2.38 (1.06) | 1.95 (0.83) | 1.47 (0.51) | 2.00 (0.53)

7. Primary Outcome: Mean Number of Inflectra Infusions at Visit 3
Time Frame: Visit 3= Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 16 | 16 | 5 | 15 | 30 | 5
infusions | 1.56 (0.63) | 1.38 (0.62) | 2.20 (1.30) | 1.47 (0.83) | 1.40 (0.50) | 1.40 (0.55)

8. Primary Outcome: Mean Number of Inflectra Infusions at Visit 4
Time Frame: Visit 4= Day 365
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: infusions
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 9 | 15 | 2 | 9 | 26 | 4
infusions | 2.56 (0.88) | 3.00 (0.85) | 2.50 (2.12) | 3.11 (1.36) | 3.08 (0.89) | 2.75 (1.71)

9. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire for Absenteeism Score at Visit 2, 3 and 4
Description: WPAI: participant rated questionnaire to determine the degree to which UC and CD affected work productivity while at work and affected activities outside of work. The scores/outcomes derived are: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism) and daily regular activity impairment. All outcomes are expressed as impairment percentages on a score range of 0 (no impairment) to 100 (maximum impairment), higher scores indicating greater impairment and less productivity.
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: The full analysis set included all participants who signed the informed consent and met the study inclusion/exclusion criteria in the study design, or the subgroups as following: those who newly initiated Inflectra, transitioned to Inflectra from Remicade or switched to Inflectra from other biologics. Here 'number analyzed' signifies participants evaluable for each specified category.
Measure: Mean (Standard Error); unit: percentage of work time missed
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
percentage of work time missed
  Change at Visit 2: number analyzed (Participants) | 9 | 13 | 2 | 11 | 25 | 7
  Change at Visit 2 | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -3.68 (2.61) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 3: number analyzed (Participants) | 12 | 12 | 3 | 10 | 26 | 3
  Change at Visit 3 | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -2.04 (2.36) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 4: number analyzed (Participants) | 10 | 13 | 3 | 9 | 22 | 3
  Change at Visit 4 | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -5.42 (2.62) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.

10. Secondary Outcome: Change From Baseline in WPAI Questionnaire for Presenteeism Score at Visit 2, 3 and 4
Description: as for outcome 9
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: percentage of impairment
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
percentage of impairment
  Change at Visit 2: number analyzed (Participants) | 10 | 13 | 2 | 11 | 25 | 7
  Change at Visit 2 | -23.7 (12) | -13.18 (6) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 3.91 (3.91) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 3: number analyzed (Participants) | 11 | 12 | 3 | 10 | 26 | 4
  Change at Visit 3 | -33.85 (11.34) | -13.53 (6.5) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 1.02 (4.07) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 4: number analyzed (Participants) | 10 | 13 | 2 | 9 | 22 | 3
  Change at Visit 4 | -39.94 (11.16) | -17.76 (5.79) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -2.14 (4.1) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.

11. Secondary Outcome: Change From Baseline in WPAI Questionnaire for Overall Work Impairment Score at Visit 2, 3 and 4
Description: as for outcome 9
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: percentage of overall work impairment
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
percentage of overall work impairment
  Change at Visit 2: number analyzed (Participants) | 9 | 13 | 2 | 11 | 25 | 7
  Change at Visit 2 | -22.21 (11.54) | -14.39 (5.88) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 2.33 (4.7) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 3: number analyzed (Participants) | 11 | 12 | 3 | 10 | 26 | 3
  Change at Visit 3 | -30.2 (10.16) | -14.93 (6.5) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 0.27 (4.65) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 4: number analyzed (Participants) | 10 | 13 | 3 | 8 | 22 | 3
  Change at Visit 4 | -38.28 (10.02) | -18.82 (5.82) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -4.8 (4.52) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.

12. Secondary Outcome: Change From Baseline in WPAI Questionnaire for Daily Regular Activity Impairment Score at Visit 2, 3 and 4
Description: as for outcome 9
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: percentage of daily activity impairment
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
percentage of daily activity impairment
  Change at Visit 2: number analyzed (Participants) | 17 | 18 | 6 | 20 | 36 | 9
  Change at Visit 2 | -35.51 (7.92) | -14.66 (4.39) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -17.27 (6.05) | 3.75 (3.92) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 3: number analyzed (Participants) | 16 | 16 | 6 | 16 | 33 | 5
  Change at Visit 3 | -43.33 (7.66) | -12.73 (6.14) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -14.09 (6.39) | -0.86 (4.59) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 4: number analyzed (Participants) | 12 | 17 | 4 | 13 | 29 | 5
  Change at Visit 4 | -46.11 (8.36) | -18.06 (6.26) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -27.64 (6.39) | -2.84 (6.1) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.

13. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication Version II (TSQM vII) for Convenience Score at Visit 2, 3 and 4
Description: TSQM vII was used to assess experiences of participants with medication on 3 dimensions: convenience, effectiveness and side effects. Convenience score utilized items 7 and 8. Items 7 and 8 were scored on the following scale: 1= extremely dissatisfied, 2= very dissatisfied, 3= dissatisfied, 4= somewhat satisfied, 5= satisfied, 6= very satisfied, 7= extremely satisfied. Convenience score was calculated using formula = ([Sum of Item 7 + Item 8] - 2)/12*100. Convenience score ranged from 0 (no convenience) to 100 (best level of convenience). Higher convenience scores indicated more convenience with medication and greater satisfaction.
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
units on a scale
  Change at Visit 2: number analyzed (Participants) | 17 | 18 | 8 | 20 | 36 | 9
  Change at Visit 2 | 7.08 (4.14) | -0.16 (4.12) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 0.75 (2.77) | 0.57 (2.91) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 3: number analyzed (Participants) | 17 | 15 | 6 | 16 | 33 | 6
  Change at Visit 3 | 6.77 (4.42) | 4.55 (5.38) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -4.01 (4.66) | 3.65 (3.1) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 4: number analyzed (Participants) | 12 | 17 | 4 | 13 | 30 | 5
  Change at Visit 4 | 8.37 (5.87) | 4.53 (5.59) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -1.44 (3.95) | -1.45 (2.97) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.

14. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication Version II (TSQM vII) for Effectiveness Score at Visit 2, 3 and 4
Description: TSQM vII was used to assess experiences of participants with medication on 3 dimensions: convenience, effectiveness and side effects. Effectiveness score utilized items 1 and 2. Items 1 and 2 were scored on the following scale: 1= extremely dissatisfied, 2= very dissatisfied, 3= dissatisfied, 4= somewhat satisfied, 5= satisfied, 6= very satisfied, 7= extremely satisfied. Effectiveness score was calculated using formula= ([Sum of Item 1 + Item 2] - 2)/12*100. Effectiveness score ranged from 0 (not effective) to 100 (highest level of effectiveness). Higher effectiveness scores indicated medication was more effective and greater satisfaction.
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
units on a scale
  Change at Visit 2: number analyzed (Participants) | 17 | 17 | 8 | 20 | 36 | 9
  Change at Visit 2 | 23.33 (6.65) | 3.27 (4.75) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 12.55 (5.25) | -10.73 (4.7) | 12.44 (9.98)
  Change at Visit 3: number analyzed (Participants) | 17 | 15 | 6 | 16 | 34 | 6
  Change at Visit 3 | 24.19 (6.88) | 10.27 (5.27) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 14.16 (7.54) | -6.66 (4.48) | 11.98 (11.77)
  Change at Visit 4: number analyzed (Participants) | 12 | 17 | 4 | 13 | 29 | 5
  Change at Visit 4 | 28.54 (8.55) | 12.95 (5.14) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 24.45 (5.98) | -4.97 (5.39) | -5.72 (19.65)

15. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication Version II (TSQM vII) for Side Effects Score at Visit 2, 3 and 4
Description: TSQM vII was used to assess experiences of participants with medication on 3 dimensions: convenience, effectiveness and side effects. Side effects score utilized items 4, 5 and 6. Items 4, 5 and 6 were scored on the following scale: 1= extremely dissatisfied, 2= very dissatisfied, 3= somewhat dissatisfied, 4= slightly dissatisfied, 5= not at all dissatisfied. Side effects score was calculated using formula = ([Sum of Item 4 + Item 5 + Item 6] - 3)/12*100, if one item is missing then: ([Sum of two completed items from 4 to 6] - 2]/8*100. Side effects score ranged from 0 (maximum side effects) to 100 (no side effects). Higher side effects scores indicated less side effects with medication and greater satisfaction.
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
units on a scale
  Change at Visit 2: number analyzed (Participants) | 10 | 13 | 6 | 13 | 24 | 4
  Change at Visit 2 | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 1.23 (2.96) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 15.32 (5.12) | -1.19 (6.23) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 3: number analyzed (Participants) | 11 | 7 | 4 | 8 | 24 | 3
  Change at Visit 3 | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 1.46 (4.25) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 13.34 (3.86) | -0.3 (5.85) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.
  Change at Visit 4: number analyzed (Participants) | 9 | 8 | 2 | 7 | 22 | 4
  Change at Visit 4 | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | -5.49 (4.25) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 15.15 (5.52) | 2.93 (5.27) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report.

16. Secondary Outcome: Mean of Total Number of Hospitalizations at Visit 1, 2, 3 and 4
Description: In this outcome measure mean of total number of hospitalizations at specified time points as a part of healthcare resource utilization assessment are reported.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hospitalization visits
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
hospitalization visits
  Visit 1 | 0.17 (0.38) | 0.00 (0.00) | 0.33 (0.71) | 0.24 (0.54) | 0.00 (0.00) | 0.40 (0.52)
  Visit 2: number analyzed (Participants) | 17 | 19 | 8 | 20 | 36 | 9
  Visit 2 | 0.06 (0.24) | 0.00 (0.00) | 0.00 (0.00) | 0.05 (0.22) | 0.17 (0.51) | 0.22 (0.67)
  Visit 3: number analyzed (Participants) | 17 | 18 | 6 | 16 | 36 | 6
  Visit 3 | 0.00 (0.00) | 0.06 (0.24) | 0.17 (0.41) | 0.06 (0.25) | 0.00 (0.00) | 0.00 (0.00)
  Visit 4: number analyzed (Participants) | 12 | 18 | 4 | 13 | 32 | 5
  Visit 4 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.08 (0.28) | 0.03 (0.18) | 0.40 (0.89)

17. Secondary Outcome: Mean of Total Number of Overall Emergency Department (ED) Visits at Visit 1, 2, 3 and 4
Description: In this outcome measure mean of total number of ED visits at specified time points as a part of healthcare resource utilization assessment are reported.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: emergency department visits
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
emergency department visits
  Visit 1 | 0.22 (0.43) | 0.10 (0.44) | 0.11 (0.33) | 0.14 (0.36) | 0.03 (0.17) | 0.20 (0.42)
  Visit 2: number analyzed (Participants) | 17 | 19 | 8 | 20 | 36 | 9
  Visit 2 | 0.06 (0.24) | 0.05 (0.23) | 0.25 (0.71) | 0.35 (1.35) | 0.11 (0.40) | 0.00 (0.00)
  Visit 3: number analyzed (Participants) | 17 | 18 | 6 | 16 | 36 | 6
  Visit 3 | 0.06 (0.24) | 0.00 (0.00) | 0.00 (0.00) | 0.06 (0.25) | 0.03 (0.17) | 0.00 (0.00)
  Visit 4: number analyzed (Participants) | 12 | 18 | 4 | 13 | 32 | 5
  Visit 4 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.09 (0.53) | 0.80 (1.10)

18. Secondary Outcome: Mean of Total Number of Outpatient Visits at Visit 1, 2, 3 and 4
Description: In this outcome measure mean of total number of outpatient visits at specified time points as a part of healthcare resource utilization assessment are reported.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: outpatient visits
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
outpatient visits
  Visit 1 | 2.06 (5.34) | 1.10 (1.95) | 4.22 (7.51) | 1.05 (1.56) | 0.78 (1.55) | 1.80 (3.49)
  Visit 2: number analyzed (Participants) | 17 | 19 | 8 | 20 | 36 | 9
  Visit 2 | 1.41 (1.33) | 1.37 (1.42) | 1.38 (1.30) | 1.60 (1.54) | 1.33 (1.39) | 1.44 (1.13)
  Visit 3: number analyzed (Participants) | 17 | 18 | 6 | 16 | 36 | 6
  Visit 3 | 1.18 (1.33) | 0.61 (0.98) | 2.50 (3.21) | 1.56 (1.15) | 0.97 (1.54) | 1.00 (0.89)
  Visit 4: number analyzed (Participants) | 12 | 18 | 4 | 13 | 32 | 5
  Visit 4 | 1.08 (1.16) | 1.33 (1.33) | 3.00 (1.41) | 1.31 (1.18) | 1.47 (1.50) | 3.40 (3.91)

19. Secondary Outcome: Mean of Total Number of Gastroenterology (GE) Outpatient Visits at Visit 1, 2, 3 and 4
Description: In this outcome measure mean of total number of gastroenterology outpatient visits at specified time points as a part of healthcare resource utilization assessment are reported.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: GE outpatient visits
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
GE outpatient visits
  Visit 1 | 0.94 (1.76) | 0.48 (0.60) | 2.67 (4.03) | 0.90 (1.45) | 0.28 (0.74) | 1.00 (1.63)
  Visit 2: number analyzed (Participants) | 17 | 19 | 8 | 20 | 36 | 9
  Visit 2 | 0.76 (0.75) | 0.42 (0.51) | 0.50 (0.76) | 0.70 (0.73) | 0.47 (0.70) | 1.11 (0.78)
  Visit 3: number analyzed (Participants) | 17 | 18 | 6 | 16 | 36 | 6
  Visit 3 | 0.59 (0.62) | 0.22 (0.43) | 0.67 (1.21) | 1.00 (0.97) | 0.36 (0.68) | 0.67 (0.52)
  Visit 4: number analyzed (Participants) | 12 | 18 | 4 | 13 | 32 | 5
  Visit 4 | 0.58 (0.79) | 0.61 (0.70) | 0.75 (0.50) | 0.62 (0.65) | 0.72 (0.89) | 1.20 (0.84)

20. Secondary Outcome: Mean of Total Number of General Practitioner (GP) Outpatient Visits at Visit 1, 2, 3 and 4
Description: In this outcome measure mean of total number of general practitioner outpatient visits at specified time points as a part of healthcare resource utilization assessment are reported.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: GP outpatient visits
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
GP outpatient visits
  Visit 1 | 0.33 (0.84) | 0.33 (0.80) | 1.33 (3.64) | 0.05 (0.22) | 0.22 (0.54) | 0.10 (0.32)
  Visit 2: number analyzed (Participants) | 17 | 19 | 8 | 20 | 36 | 9
  Visit 2 | 0.41 (0.51) | 0.63 (0.76) | 0.50 (0.76) | 0.65 (0.93) | 0.64 (0.96) | 0.22 (0.44)
  Visit 3: number analyzed (Participants) | 17 | 18 | 6 | 16 | 36 | 6
  Visit 3 | 0.29 (0.47) | 0.17 (0.38) | 1.00 (1.26) | 0.25 (0.45) | 0.33 (0.59) | 0.33 (0.52)
  Visit 4: number analyzed (Participants) | 12 | 18 | 4 | 13 | 32 | 5
  Visit 4 | 0.42 (0.67) | 0.56 (0.86) | 1.50 (1.29) | 0.46 (0.78) | 0.38 (0.75) | 1.40 (2.07)

21. Secondary Outcome: Number of Participants With Crohn's Disease Remission at Visit 1, 2, 3 and 4
Description: Participants with a confirmed diagnosis of CD, were said to have remission when Harvey-Bradshaw index (HBI) score was less than (<) 5. HBI measures 5 parameters; the general well-being (0= very well to 4= terrible), abdominal pain (0= none to 3= severe), number of liquid stools per day (0 to no maximum score), presence of an abdominal mass on physical exam (0= none to 3= definite and tender), and whether there are any complications (0= no complications, 1= arthralgia, 2= uveitis, 3= erythema nodosum, 4= aphthous ulcer, 5= pyoderma gangrenosum, 6= anal fissure, 7= new fistula, 8= abscess). The total HBI score: sum of all the 5 individual parameters, the minimum score is 0 and there was no pre-specified maximum score as it depended on the number of liquids stools. Higher HBI scores = greater disease activity.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 21 | 36 | 10
Participants
  Visit 1 | 13 | 28 | 7
  Visit 2: number analyzed (Participants) | 20 | 36 | 9
  Visit 2 | 16 | 23 | 8
  Visit 3: number analyzed (Participants) | 16 | 36 | 6
  Visit 3 | 12 | 24 | 3
  Visit 4: number analyzed (Participants) | 13 | 32 | 5
  Visit 4 | 11 | 23 | 3

22. Secondary Outcome: Number of Participants With Ulcerative Colitis Remission at Visit 1, 2, 3 and 4
Description: Participants with a confirmed diagnosis of UC, were said to have remission when there was a reduction of partial Mayo score (PMS) of <3 points from baseline. PMS comprised of 3 parameters: stool frequency (0= normal number of stools to 3= having >=5 stools more than normal), most severe rectal bleeding of the day (0= no blood seen to 3= pure blood passed), and physician's global assessment (0= normal to 3= severe disease). The total PMS was the sum of all the parameters, score ranging from 0 (normal or inactive disease) to 9 (severe disease). Higher scores indicated more severe disease.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9
Participants
  Visit 1 | 1 | 15 | 1
  Visit 2: number analyzed (Participants) | 17 | 19 | 8
  Visit 2 | 14 | 16 | 4
  Visit 3: number analyzed (Participants) | 17 | 18 | 6
  Visit 3 | 12 | 14 | 3
  Visit 4: number analyzed (Participants) | 12 | 18 | 4
  Visit 4 | 10 | 16 | 1

23. Secondary Outcome: Number of Participants With Crohn's Disease Response at Visit 1, 2, 3 and 4
Description: Participants with a confirmed diagnosis of CD, were said to have response when there was reduction of HBI score of >=3 points from baseline. HBI measures 5 parameters; the general well-being (0= very well to 4= terrible), abdominal pain (0= none to 3= severe), number of liquid stools per day (0 to no maximum score), presence of an abdominal mass on physical exam (0= none to 3= definite and tender), and whether there are any complications (0= no complications, 1= arthralgia, 2= uveitis, 3= erythema nodosum, 4= aphthous ulcer, 5= pyoderma gangrenosum, 6= anal fissure, 7= new fistula, 8= abscess). The total HBI score: sum of all the 5 individual parameters, the minimum score is 0 and there was no pre-specified maximum score as it depended on the number of liquids stools. Higher HBI scores = greater disease activity.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 21 | 36 | 10
Participants
  Visit 1 | 0 | 0 | 0
  Visit 2: number analyzed (Participants) | 20 | 36 | 9
  Visit 2 | 4 | 3 | 3
  Visit 3: number analyzed (Participants) | 16 | 36 | 6
  Visit 3 | 5 | 4 | 2
  Visit 4: number analyzed (Participants) | 13 | 32 | 5
  Visit 4 | 4 | 2 | 1

24. Secondary Outcome: Number of Participants With Ulcerative Colitis Response at Visit 1, 2, 3 and 4
Description: Participants with a confirmed diagnosis of UC, were said to have response when there was a reduction of partial Mayo score of >=3 points from baseline. PMS comprised of 3 parameters: stool frequency (0= normal number of stools to 3= having >=5 stools more than normal), most severe rectal bleeding of the day (0= no blood seen to 3= pure blood passed), and physician's global assessment (0= normal to 3= severe disease). The total PMS was the sum of all the parameters, score ranging from 0 (normal or inactive disease) to 9 (severe disease). Higher scores indicated more severe disease.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9
Participants
  Visit 1 | 0 | 0 | 0
  Visit 2: number analyzed (Participants) | 17 | 19 | 8
  Visit 2 | 12 | 2 | 4
  Visit 3: number analyzed (Participants) | 17 | 18 | 6
  Visit 3 | 13 | 2 | 3
  Visit 4: number analyzed (Participants) | 12 | 18 | 4
  Visit 4 | 8 | 2 | 2

25. Secondary Outcome: Change From Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) at Visit 2, 3 and 4
Description: This questionnaire is designed to find out how participants felt during the last 2 weeks. Participants were asked 10 questions about physical, social, and emotional status. Participants had to respond for every question on a scale from 1 (poor) to 7 (good). Total SIBDQ score was sum of scores from 10 questions, with range from 10 (poor quality of life) to 70 (optimum quality of life), higher values indicated better well-being.
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
units on a scale
  Change at Visit 2: number analyzed (Participants) | 17 | 18 | 8 | 20 | 36 | 9
  Change at Visit 2 | 17.52 (3.13) | 4.96 (2.2) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 6.73 (2.34) | -0.19 (1.19) | 12.72 (6.19)
  Change at Visit 3: number analyzed (Participants) | 17 | 16 | 6 | 16 | 35 | 6
  Change at Visit 3 | 21.23 (3.48) | 6.4 (1.97) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 7.71 (2.88) | 0.46 (1.22) | 11.97 (5.41)
  Change at Visit 4: number analyzed (Participants) | 12 | 17 | 4 | 13 | 30 | 5
  Change at Visit 4 | 23.57 (3.9) | 8.29 (2.6) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 9.7 (2.62) | 0.86 (1.75) | 11.7 (1.57)

26. Secondary Outcome: Change From Baseline in Quality of Life Visual Analog Scale (VAS) at Visit 2, 3 and 4
Description: Participants were asked to mark their overall well-being at specified visits on a scale from 0 millimeter to 100 millimeter. 0 indicated worst health and 100 indicated perfect health. Higher scores indicated better well-being.
Time Frame: Baseline (before initiation of Inflectra); Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 9
Measure: Mean (Standard Error); unit: millimeter
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
millimeter
  Change at Visit 2: number analyzed (Participants) | 17 | 18 | 8 | 20 | 36 | 9
  Change at Visit 2 | 16.68 (4.12) | 2.31 (2.41) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 6.16 (5.97) | 0.67 (2.79) | 6.83 (6.52)
  Change at Visit 3: number analyzed (Participants) | 17 | 16 | 6 | 16 | 35 | 6
  Change at Visit 3 | 17.93 (4.28) | 6.49 (2.23) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 6.75 (5.88) | 0.23 (2.38) | 4.89 (7.44)
  Change at Visit 4: number analyzed (Participants) | 12 | 17 | 4 | 13 | 30 | 5
  Change at Visit 4 | 13.6 (5.25) | 9.88 (3.31) | NA (NA) — Data could not be calculated as statistical model did not converge, hence no results available to report. | 13.56 (6.11) | 1.75 (1.74) | 1.22 (12.63)

27. Secondary Outcome: Number of Participants Categorized on the Basis of Montreal Classification by Extent: Ulcerative Colitis
Description: Participants with Montreal classification for UC were reported for extent (E1 ulcerative proctitis, E2 left-sided UC, E3 extensive UC, unknown).
Time Frame: Baseline (before initiation of Inflectra)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9
Participants
  E1 Ulcerative proctitis | 3 | 1 | 1
  E2 Left-sided UC | 6 | 3 | 4
  E3 Extensive UC | 8 | 16 | 4
  Unknown | 1 | 1 | 0

28. Secondary Outcome: Number of Participants Categorized on the Basis of Montreal Classification by Location and Behavior: Crohn's Disease
Description: Participants with Montreal classification for CD was reported for behavior (B1: nonstricturing, no penetrating, B2: structuring, B3: penetrating, P: perianal disease, unknown) and location (L1: terminal ileum, L2: colon, L3: ileocolon, L4: upper gastrointestinal [GI]).
Time Frame: Baseline (before initiation of Inflectra)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 21 | 36 | 10
Participants
  Location: L1 Terminal ileum | 7 | 12 | 3
  Location: L2 Colon | 6 | 12 | 4
  Location: L3 Ileocolon | 8 | 7 | 3
  Location: L4 Upper GI | 0 | 1 | 0
  Location: Unknown | 0 | 4 | 0
  Behavior: B1 Nonstricturing, nonpenetrating | 11 | 3 | 6
  Behavior: B2 Stricturing | 4 | 6 | 1
  Behavior: B3 Penetrating | 4 | 0 | 1
  Behavior: P Perianal disease | 0 | 2 | 1
  Behavior: Unknown | 2 | 25 | 1

29. Secondary Outcome: Partial Mayo Score (PMS) at Baseline for Participants With Ulcerative Colitis
Description: PMS comprised of 3 parameters: stool frequency (0= normal number of stools to 3= having >=5 stools more than normal), most severe rectal bleeding of the day (0= no blood seen to 3= pure blood passed), and physician's global assessment (0= normal to 3= severe disease). The total PMS was the sum of all the parameters, score ranging from 0 (normal or inactive disease) to 9 (severe disease). Higher scores indicated more severe disease.
Time Frame: Baseline (before initiation of Inflectra)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9
units on a scale | 5.67 (2.25) | 1.38 (1.83) | 6.00 (2.65)

30. Secondary Outcome: Harvey Bradshaw Index (HBI) at Baseline for Participants With Crohn's Disease
Description: HBI measures 5 parameters; the general well-being (0= very well to 4= terrible), abdominal pain (0= none to 3= severe), number of liquid stools per day (0 to no maximum score), presence of an abdominal mass on physical exam (0= none to 3= definite and tender), and whether there are any complications (0= no complications, 1= arthralgia, 2= uveitis, 3= erythema nodosum, 4= aphthous ulcer, 5= pyoderma gangrenosum, 6= anal fissure, 7= new fistula, 8= abscess). The total HBI score: sum of all the 5 individual parameters, the minimum score is 0 and there was no pre-specified maximum score as it depends depended on the number of liquids stools. Higher HBI scores = greater disease activity.
Time Frame: Baseline (before initiation of Inflectra)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 21 | 36 | 10
units on a scale | 3.95 (3.15) | 3.11 (3.05) | 3.57 (2.51)

31. Secondary Outcome: Number of Participants With Infections
Description: In this outcome measure, number of participants who had infections as adverse events are reported under 2 categories: 1) all infections (including both serious and non-serious adverse events) and 2) serious infections (serious adverse event). An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect.
Time Frame: Visit 1 to 4 (approximately 1 year)
Population: The safety analysis set included all participants who signed an informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
Participants
  All Infections | 0 | 1 | 0 | 0 | 0 | 0
  Serious Infections | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Number of Participants With Malignancy and Lymphoma
Description: In this outcome measure, number of participants who had malignancy and lymphoma as adverse events are reported under 2 categories: 1) malignancy and lymphoma (serious adverse event) and 2) malignancy and lymphoma (non-serious adverse event. An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect.
Time Frame: Visit 1 to 4 (approximately 1 year)
Population: The safety analysis set included all participants who signed an informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
Participants
  Malignancy and Lymphoma (Serious Adverse Event) | 0 | 0 | 0 | 0 | 3 | 0
  Malignancy and Lymphoma (Non-serious Adverse Event) | 0 | 0 | 0 | 1 | 0 | 0

33. Secondary Outcome: Number of Participants With Infusion-related Reactions
Description: In this outcome measure, number of participants who had infusion-related reactions as adverse events are reported under 2 categories: 1) infusion-related reactions (serious adverse event) and 2) infusion-related reactions (non-serious adverse event) are reported. An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect.
Time Frame: Visit 1 to 4 (approximately 1 year)
Population: The safety analysis set included all participants who signed an informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
Participants
  Infusion-related reactions (serious adverse event) | 0 | 0 | 0 | 0 | 0 | 0
  Infusion-related reactions (non-serious adverse event) | 1 | 1 | 0 | 0 | 0 | 0

34. Secondary Outcome: Number of Participants With Any Serious Adverse Event
Description: An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect.
Time Frame: Visit 1 to 4 (approximately 1 year)
Population: The safety analysis set included all participants who signed an informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
Participants | 0 | 3 | 1 | 5 | 8 | 2

35. Other Pre Specified Outcome: Duration of Inflectra Therapy
Description: In this outcome measure duration of Inflectra treatment (in months) is reported.
Time Frame: Visit 1 to 4 (approximately 1 year)
Population: The safety analysis set included all participants who signed an informed consent. Here "Overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 35 | 10
months | 11.13 (3.71) | 10.42 (3.67) | 8.90 (4.40) | 10.37 (3.22) | 11.83 (2.27) | 9.59 (3.70)

36. Other Pre Specified Outcome: Number of Participants With Any Changes in Dosing
Description: In this outcome measure, number of participants who had any changes in dosing are reported.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: The safety analysis set included all participants who signed an informed consent. Here 'number analyzed' signifies participants evaluable for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
Participants
  Visit 1 | 3 | 5 | 0 | 1 | 7 | 1
  Visit 2: number analyzed (Participants) | 17 | 19 | 8 | 20 | 36 | 9
  Visit 2 | 6 | 4 | 4 | 10 | 1 | 4
  Visit 3: number analyzed (Participants) | 17 | 18 | 6 | 16 | 36 | 6
  Visit 3 | 5 | 2 | 2 | 3 | 3 | 1
  Visit 4: number analyzed (Participants) | 12 | 18 | 4 | 13 | 32 | 5
  Visit 4 | 3 | 2 | 1 | 6 | 4 | 2

37. Other Pre Specified Outcome: Number of Participants Who Completed Each Study Visit
Description: In this outcome measure, number of participants who completed specified study visits are reported as evaluation of treatment adherence.
Time Frame: Visit 1= Day 1; Visit 2= Day 90; Visit 3= Day 180; Visit 4= Day 365
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
Number analyzed (Participants) | 18 | 21 | 9 | 21 | 36 | 10
Participants
  Visit 1 | 18 | 21 | 9 | 21 | 36 | 10
  Visit 2 | 17 | 19 | 8 | 20 | 36 | 9
  Visit 3 | 17 | 18 | 6 | 16 | 36 | 6
  Visit 4 | 12 | 18 | 4 | 13 | 32 | 5

ADVERSE EVENTS:
Time Frame: Visit 1 to 4 (approximately 1 year)
Description: Same event may appear as both an AE and Serious Adverse Events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety set.
Arm/Group | UC: New Inflectra | UC: Inflectra After Remicade | UC: Inflectra After Other Biologics | CD: New Inflectra | CD: Inflectra After Remicade | CD: Inflectra After Other Biologics
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21 | 0/9 | 0/21 | 0/36 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/18 | 3/21 | 1/9 | 5/21 | 8/36 | 2/10
Other Adverse Events (participants affected / at risk) | 2/18 | 4/21 | 5/9 | 6/21 | 7/36 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UC: New Inflectra (N=18) | UC: Inflectra After Remicade (N=21) | UC: Inflectra After Other Biologics (N=9) | CD: New Inflectra (N=21) | CD: Inflectra After Remicade (N=36) | CD: Inflectra After Other Biologics (N=10)
Abdominal abscess (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colon stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Colovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Small bowel obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Drug ineffective (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Liver abscess (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug specific antibody present (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Near syncope during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UC: New Inflectra (N=18) | UC: Inflectra After Remicade (N=21) | UC: Inflectra After Other Biologics (N=9) | CD: New Inflectra (N=21) | CD: Inflectra After Remicade (N=36) | CD: Inflectra After Other Biologics (N=10)
Thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative aggravated (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Disease recurrence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Perianal abscess (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzymes increased (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteoporosis/osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Low-grade B cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT03801928/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT03801928/SAP_001.pdf